CLINICAL TRIAL: NCT06178965
Title: Incisional Hernia Repair by Abdominal Wall Component Release With Contemporary Onlay Mesh Fixation
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Zagazig University (Other Government)
Responsible Party: Principal Investigator, Yasser Ali Orban, assisstant professor, Zagazig University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: incisional hernia repair
Record Dates: First submitted 2023-12-16; First posted 2023-12-21 (Actual); Last update posted 2023-12-21 (Actual); Status verified 2023-12

CONDITIONS: Incisional Hernia; Onlay Mesh; Abdominal Wall Component Release
MeSH Terms: conditions — Incisional Hernia

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Abdominal Wall Component Release with Contemporary Onlay Mesh Fixation (Other): Abdominal Wall Component Release with Contemporary Onlay Mesh Fixation in patients with incisional hernia
  Interventions: Procedure: Incisional Hernia Repair by Abdominal Wall Component Release with Contemporary Onlay Mesh Fixation

INTERVENTIONS:
Procedure: Incisional Hernia Repair by Abdominal Wall Component Release with Contemporary Onlay Mesh Fixation — patients with incisional hernia will be operated by hernia reduction and sac closure followed by placement of onlay mesh after creating suitable flaps.

SUMMARY:
There is a great expansion in the presentation of complex incisional hernia defects. Primary closure for most cases is impossible with a high rate of recurrence. Component separation provides an autologous repair of the defect but still has considerable recurrence rate. Reinforcement of component separation provides a more strength full repair and may be less recurrence.

DETAILED DESCRIPTION:
the surgical correction was done under general anesthesia. After scrubbing and draping, an elliptical incision was performed .

Open the hernia sac then reduce the contents with adhesolysis as required. subcutaneous flaps on both sides were created in a manner that permit to spread an 8 cm mesh after the closure of the abdominal wall. approximate the facia after trimming of its edges with clamps with a manner that allow 1to 2 cm overlap in the midline without tension.

In case of tension do selective myofascial advancement (sequential components release). Our steps would be first a unilateral posterior rectus sheath release (1-2 cm longuitodinal incision lateral to linea alba) and reassess, if tension still present, bilateral posterior sheath release should be performed.If tension still present, do a unilateral then bilateral external oblique release as required (1-2 cm lateral to the linea semilunaris along the length of the abdominal wall).

close the defect with prolene 1 then cover with onlay wide pore mesh fixation with 2/0 prolene. Close the skin after placement of 2 subcutaneous suction drains.

ELIGIBILITY:
Inclusion Criteria:

* Age of 16 years and older.
* Both sexes.
* Patients with clean incisional hernia of stage I, II and III according to the ventral hernia staging system were included.

Exclusion Criteria:

* - Obese patients with BMI ≥35 kg/m2, Patients with contaminated hernia stage II and III, patients with collagen disease, patients with history of aortobifemoral bypass, Patients refusing mesh hernioplasty, Females in childbearing age who looks for further children, Patients unfit for surgery according to ASA criteria, Patients with a parastomal hernia, patient with a stoma and patients with uncontrolled diabetics, active smokers, and patients with COPD were excluded

Min Age: 16 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-12-01 (Actual); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
detect black color at the incision site | postoperative day 1 and 2
  the detection by vision

SECONDARY OUTCOMES:
detect pulge at incision site | from postoperative day 1 to 6 months postoperative
  detect by vision

CONTACTS AND LOCATIONS:
Locations (1):
- Zagazig University, Zagazig, Egypt